CLINICAL TRIAL: NCT00502307
Title: A Phase 2, Placebo-Controlled, Randomized, Discontinuation Trial of Tivozanib (AV-951) in Patients With Renal Cell Carcinoma
Brief Title: A Study of Tivozanib (AV-951), an Oral VEGF Receptor Tyrosine Kinase Inhibitor, in the Treatment of Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AV-951-07-201
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Results first posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal Cell Carcinoma; AV-951; tivozanib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tivozanib (AV-951) administered as a solid dosage form daily for three weeks per month
  Interventions: Drug: Tivozanib (AV-951)
- 2 (Placebo Comparator): solid oral capsule containing excipients dosed daily for three weeks per month
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Tivozanib (AV-951) — solid oral dosage form taken daily for three weeks per one month cycle
  Arms: 1
Drug: Placebo comparator — solid oral capsule containing excipients dosed daily for three weeks per month
  Arms: 2

SUMMARY:
This phase 2 trial is evaluating the antineoplastic activity of tivozanib (AV-951) in treating patients with recurrent or metastatic renal cell cancer. Tivozanib (AV-951) is a VEGF-receptor tyrosine kinase inhibitor, and may stop the growth of tumor cells by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
Approximately 200 patients will be enroled into the initial, 16 week, open-label period using 1.5 mg/day dosing. Patients will receive tivozanib (AV-951) continuously for 3 weeks followed by 1 week off study drug. Patients will undergo disease assessment at baseline and after Cycles 2 and 4 and response will be determined by RESIST criteria.

After the initial, 16 week open-label period, disease status will be assessed and compared to baseline using modified RECIST criteria:

* Patients with greater than or equal to 25% tumor shrinkage will continue on their current dose of tivozanib (AV-951)
* Patients with less than 25% tumor change (growth or shrinkage) will be randomly assigned to double-blind tivozanib (AV-951) or matching placebo for 12 weeks
* Patients with greater than or equal to 25% tumor growth will be discontinued

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 year old males or females
* Patients with recurrent or metastatic renal cell carcinoma (RCC) or primary RCC that is not amendable to surgical intervention
* Histologically or cytologically confirmed renal cell carcinoma
* Measurable disease
* No more than one prior systemic treatment (chemotherapy or immunotherapy) for RCC.
* No active brain metastases
* Karnofsky performance status ≥ 70%, life expectancy ≥ 3 months
* No childbearing potential, or use of effective contraception during the study and for 4 weeks after the last dose of study drug
* Archival paraffin embedded tumor tissue, if available.
* Ability to give written informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Primary CNS malignancies; active CNS metastases
* Hematologic malignancies (includes: leukemia, any form; lymphoma; and multiple myeloma)
* Any of the following hematologic abnormalities:

  * Hemoglobin ≤ 9.0 g/dL
  * ANC < 1500 per mm3
  * Platelet count < 100,000 per mm3
* Any of the following serum chemistry abnormalities:

  * Total bilirubin > 1.5 × the ULN
  * AST or ALT ≥ 2.5 × the ULN
  * Serum albumin < 3.0 g/dL
  * Creatinine > 1.7 × ULN (or calculated CLCR <50 mL/min/1.73 m2)
  * Proteinuria > 2.5 g/24 hours or 4+ with urine dipstick
* Significant cardiovascular disease, including:

  * Active clinically symptomatic left ventricular failure
  * Active HTN (diastolic blood pressure > 100 mmHg). Patients with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 4 weeks
  * Uncontrolled hypertension: Blood pressure >140/90 mmHg on more than 2 antihypertensive medications.
  * Myocardial infarction within 3 months prior to administration of first study dose
* Unhealed wounds (including active gastric ulcers)
* Serious/active infection; infection requiring parenteral antibiotics
* Inadequate recovery from prior antineoplastic therapy
* Inadequate recovery from any prior surgical procedure; major surgical procedure within 4 weeks prior to study entry
* Life-threatening illness or organ system dysfunction compromising safety evaluation
* Psychiatric disorder, altered mental status precluding informed consent or necessary testing
* Inability to comply with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy G Nosov, M.D., Principal Investigator — Russian Oncological Research Center n.a. N.N. Blokhin of the Russian Academy of Medical Sciences
Locations (24):
- India (5):
  - Vellore, Tamil Nadu
  - Kolkata
  - Mumbai
  - New Delhi
  - Pune
- Russia (12):
  - Astrakhan
  - Kazan'
  - Moscow
  - Obninsk
  - Pyatigorsk
  - Rostove-on-Don
  - Saint Petersburg
  - Sochi
  - Tomsk
  - Ufa
  - Veliky Novgorod
  - Yoshkar-Ola
- Ukraine (7):
  - Cherkassy
  - Dnipro
  - Donetsk
  - Kharkiv
  - Lviv
  - Uzhhorod
  - Zaporizzhya

REFERENCES:
- [Derived] Barata PC, Chehrazi-Raffle A, Allman KD, Asnis-Alibozek A, Kasturi V, Pal SK. Activity of Tivozanib in Non-clear Cell Renal Cell Carcinoma: Subgroup Analysis From a Phase II Randomized Discontinuation Trial. Oncologist. 2023 Oct 3;28(10):894-900. doi: 10.1093/oncolo/oyad132. PMID 37315114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all the inclusion and none of the exclusion criteria were enrolled
Pre-assignment Details: All participants underwent inclusion and exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study related procedures.
  All the study assessments were performed as per the schedule of assessment.
Groups:
- Open-label Period: Tivozanib (AV-951): Subjects were enrolled into the initial, 16-week, open-label period and received tivozanib at a dose of 1.5 mg/day (oral administration). Subjects received tivozanib continuously for 3 weeks followed by 1 week off study drug (1 cycle = 3 weeks on, 1 week off).
- Double-blind Period: Tivozanib (AV-951): Subjects with < 25% tumor change (growth or shrinkage) at the end of the 16-week open-label period were randomly assigned to receive 1.5 mg/ day of tivozanib for 12 weeks (3 cycles; 1 cycle = 3 weeks on, 1 week off) in a double-blind manner.
- Double-blind Period: Placebo: Subjects with < 25% tumor change (growth or shrinkage) at the end of the 16-week open-label period were randomly assigned to receive matching placebo for 12 weeks (3 cycles; 1 cycle = 3 weeks on, 1 week off) in a double-blind manner.
Period: Open Label Period (16 Weeks)
Arm/Group | Open-label Period: Tivozanib (AV-951) | Double-blind Period: Tivozanib (AV-951) | Double-blind Period: Placebo
Started | 272 | 0 | 0
Completed | 196 | 0 | 0
Not Completed | 76 | 0 | 0
Not completed — Progressive disease | 50 | 0 | 0
Not completed — Discontinued due to other reasons | 26 | 0 | 0
Period: Double-Blind Period (12 Weeks)
Arm/Group | Open-label Period: Tivozanib (AV-951) | Double-blind Period: Tivozanib (AV-951) | Double-blind Period: Placebo
Started | 0 | 61 | 57
Completed | 0 | 35 | 48
Not Completed | 0 | 26 | 9
Not completed — Progressive disease | 0 | 23 | 2
Not completed — Discontinued due to other reasons | 0 | 3 | 7
Period: Maintenance Period
Arm/Group | Open-label Period: Tivozanib (AV-951) | Double-blind Period: Tivozanib (AV-951) | Double-blind Period: Placebo
Started | 148 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 148 | 0 | 0
Not completed — Progressive disease | 80 | 0 | 0
Not completed — Discontinued due to other reasons | 68 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open-label Period:Tivozanib (AV-951): Subjects were enrolled into the initial, 16-week, open-label period and received tivozanib at a dose of 1.5 mg/day (oral administration). Subjects received tivozanib continuously for 3 weeks followed by 1 week off study drug (1 cycle = 3 weeks on, 1 week off). After 16 weeks (4 cycles), disease status was assessed and compared to baseline. Tivozanib was to be discontinued following disease progression or unacceptable toxicity.
Arm/Group | Open-label Period:Tivozanib (AV-951)
Number analyzed (Participants) | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 272
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 271
  Unknown or Not Reported | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs)/Serious AEs (SAEs)
Description: To determine the safety and tolerability of tivozanib (AV-951) with the protocol-specified dose schedule
Time Frame: 28 weeks after study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Period: Tivozanib (AV-951) | Double-blind Period: Tivozanib (AV-951) | Double-blind Period: Placebo
Number analyzed (Participants) | 272 | 61 | 57
Participants
  Adverse events | 215 | 31 | 32
  Serious adverse events | 16 | 2 | 3
  Grade 3 or higher adverse events | 86 | 8 | 10
  Treatment-related adverse events | 174 | 13 | 7
  Discontinuations due to adverse events | 10 | 1 | 3
  Deaths | 6 | 1 | 2

2. Primary Outcome: Objective Response [Complete Response (CR) + Partial Response (PR)] Rate at 16 Week Open-Label Period (All Treated Population)
Description: The ORR is defined as the rate of (CR+PR). Objective response rates following the 16-week, open-label period (investigator assessment and IRR assessment) were estimated per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and was assessed by magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Overall Response (OR) = CR + PR.
Time Frame: 16 weeks after study entry
Measure: Count of Participants; unit: Participants
Groups:
- Investigator Assessment; Independent Radiology Reviewer Assessment: All assessment were performed by the study Investigator and similarly for IRR.
Arm/Group | Investigator Assessment | Independent Radiology Reviewer Assessment
Number analyzed (Participants) | 272 | 272
Participants
  Complete response | 1 | 0
  Partial response | 66 | 49
Statistical Analysis 1: Comparison: Investigator Assessment; Test type: Other; Exact binomial distribution = 24.6, 95% CI 2-sided [19.6 to 30.2]
Statistical Analysis 2: Comparison: Independent Radiology Reviewer Assessment; Test type: Other; Exact binomial distribution = 18.0, 95% CI 2-sided [13.6 to 23.1]

3. Primary Outcome: Percentage of Randomly Assigned Subjects Remaining Progression Free at 12 Weeks Following Random Assignment to Tivozanib (AV-951) or Placebo
Description: Percentages of subjects remaining progression-free at 12 weeks post-randomization were compared across the 2 treatment arms in the ITT population. A Cochran-Mantel- Haenszel (CMH) test of general association was used, stratifying by country to evaluate the null hypothesis that treatment arm is not associated with subjects remaining progression-free. Non-completers were treated as failures. Progression is defined using RECIST v1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 28 weeks after study entry
Measure: Count of Participants; unit: Participants
Groups:
- Investigator Assessment (Tivozanib); Investigator Assessment (Placebo); Independent Radiology Reviewer (Tivozanib); Independent Radiology Reviewer (Placebo): All assessment were performed by the study Investigator and similarly for IRR.
Arm/Group | Investigator Assessment (Tivozanib) | Investigator Assessment (Placebo) | Independent Radiology Reviewer (Tivozanib) | Independent Radiology Reviewer (Placebo)
Number analyzed (Participants) | 61 | 57 | 61 | 57
Participants | 35 | 16 | 30 | 12
Statistical Analysis 1: Comparison: Investigator Assessment (Tivozanib) vs Investigator Assessment (Placebo); Test type: Other; p = 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Independent Radiology Reviewer (Tivozanib) vs Independent Radiology Reviewer (Placebo); Test type: Other; p = 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Subjects With Progression Free-survival (PFS) After Random Assignment (Randomized Sub-set Only) (at 12 Weeks Post Randomization )
Description: PFS after randomization in the ITT population was described using the Kaplan-Meier methodology. PFS was compared across treatment arms using the log-rank test.
Time Frame: 28 weeks from study entry
Measure: Count of Participants; unit: Participants
Groups:
- Independent Radiology Reviewer Assessment (Tivozanib); Independent Radiology Reviewer Assessment (Placebo): All assessment were performed by the study Investigator and similarly for IRR.
Arm/Group | Investigator Assessment (Tivozanib) | Investigator Assessment (Placebo) | Independent Radiology Reviewer Assessment (Tivozanib) | Independent Radiology Reviewer Assessment (Placebo)
Number analyzed (Participants) | 61 | 57 | 61 | 57
Participants
  Number of subjects with progression | 23 | 33 | 22 | 24
  Number of censored subjects | 38 | 24 | 39 | 33
Statistical Analysis 1: Comparison: Investigator Assessment (Tivozanib) vs Investigator Assessment (Placebo); Test type: Other; p = 0.005, Log Rank
Statistical Analysis 2: Comparison: Independent Radiology Reviewer Assessment (Tivozanib) vs Independent Radiology Reviewer Assessment (Placebo); Test type: Other; p = 0.129, Log Rank

5. Secondary Outcome: Overall Progression-free Survival (From Start of Treatment)
Description: Number of subjects with Overall PFS (from start of treatment) was estimated using the Kaplan-Meier methodology. Subjects randomized to receive placebo were censored at randomization. Withdrawals are also censored. An alternative analysis was conducted in which PFS for subjects randomized to receive tivozanib was weighted more heavily to compensate for the information loss from randomization of other subjects to receive placebo. Additional analyses in which withdrawal was considered a PFS event were also conducted.
Time Frame: 12 months from study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Investigator Assessment (Tivozanib) | Investigator Assessment (Placebo) | Independent Radiology Reviewer Assessment (Tivozanib) | Independent Radiology Reviewer Assessment (Placebo)
Number analyzed (Participants) | 61 | 57 | 61 | 57
Participants
  Number of subjects with progression | 47 | 33 | 36 | 24
  Number of censored subjects | 14 | 24 | 25 | 33
Statistical Analysis 1: Comparison: Investigator Assessment (Tivozanib) vs Investigator Assessment (Placebo); Test type: Other; p = 0.003, Log Rank
Statistical Analysis 2: Comparison: Independent Radiology Reviewer Assessment (Tivozanib) vs Independent Radiology Reviewer Assessment (Placebo); Test type: Other; p = 0.089, Log Rank

6. Secondary Outcome: Time to Peak Plasma Concentration (Tmax) of Tivozanib in a Subset of Subjects
Description: Tivozanib concentrations in human serum were determined. The PK population included all subjects who had taken at least 1 dose of tivozanib and whose PK profile(s) were evaluable. All subjects received 1.5 mg tivozanib (1.3397 mg free base) in Cycle 1.
Time Frame: Cycle 1, Day 1: Pre-dose and 2, 4 and 24 hours post dose; Cycle 1, Day 8: Pre-dose; Cycle 1, Day 21: Pre-dose and 2, 4, 24, 48, and 96 hours post dose; Cycle 2 (Day 1): Pre-dose
Population: The PK population had 21 subjects. However, there were subjects with missing data for both Cycle 1 Day 1 and Cycle 1 Day 21. Hence, the number of participants analyzed varies i.e, 20 for Cycle 1 Day 1 and 16 for Cycle 1 Day 21.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Tivozanib 1.5 mg: A total of 21 subjects received 1.5 mg tivozanib (1.3397 mg free base) in Cycle 1.
Arm/Group | Tivozanib 1.5 mg
Number analyzed (Participants) | 21
hours
  Cycle 1 Day 1: number analyzed (Participants) | 20
  Cycle 1 Day 1 | 7.122 (8.511)
  Cycle 1 Day 21: number analyzed (Participants) | 16
  Cycle 1 Day 21 | 3.64 (5.61)

7. Secondary Outcome: Maximum Observed Serum Concentration During a Dosing Interval at Steady State (Cmax)
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tivozanib 1.5 mg
Number analyzed (Participants) | 21
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 20
  Cycle 1 Day 1 | 15.51 (11.70)
  Cycle 1 Day 21: number analyzed (Participants) | 16
  Cycle 1 Day 21 | 94.29 (37.80)

8. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve From Zero to the Last Quantifiable Sampling Point [AUC(0→24)]
Description: as for outcome 6
Time Frame: 28 weeks from study entry
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Tivozanib 1.5 mg
Number analyzed (Participants) | 21
h*ng/mL
  Cycle 1 Day 1 | 258.2 (197.0)
  Cycle 1 Day 21 | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious treatment-emergent adverse events and treatment emergent adverse events in Safety (SAF) Population was reported.
Arm/Group | Open-label Period: Tivozanib (AV-951) | Double-blind Period: Tivozanib (AV-951) | Double-blind Period: Placebo
Serious Adverse Events (participants affected / at risk) | 16/272 | 2/61 | 3/57
Other Adverse Events (participants affected / at risk) | 215/272 | 31/61 | 32/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Period: Tivozanib (AV-951) (N=272) | Double-blind Period: Tivozanib (AV-951) (N=61) | Double-blind Period: Placebo (N=57)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (3)
Metatstatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Period: Tivozanib (AV-951) (N=272) | Double-blind Period: Tivozanib (AV-951) (N=61) | Double-blind Period: Placebo (N=57)
Asthenia (General disorders) | 32 (49) | 6 (9) | 7 (7)
Fatigue (General disorders) | 29 (45) | 2 (2) | 4 (6)
Pyrexia (General disorders) | 14 (16) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 10 (11) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 24 (40) | 4 (6) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (13) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (25) | 3 (4) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (17) | 0 (0) | 2 (2)
Gamma-glutamyl transferase increased (Investigations) | 15 (27) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (16) | 0 (0) | 0 (0)
Rash generalized (Skin and subcutaneous tissue disorders) | 9 (11) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (17) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 10 (11) | 3 (5) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 9 (12) | 2 (2) | 3 (3)
Combined Hypertension (Vascular disorders) | 114 (199) | 0 (0) | 0 (0) — Includes hypertension, blood pressure increased, essential hypertension, and hypertensive crisis
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 54 (76) | 3 (7) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 6 (7) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (20) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No